CLINICAL TRIAL: NCT07351383
Title: Comparison of Topical Cryoanethesia and Benzocaine in Pain Perception During Mandibular Nerve Block in Pediatric Patients: A Randomized Controlled Clinical Trial
Brief Title: Topical Cryoanesthesia Versus Benzocaine in Pediatric Dentistry
Acronym: No acronym
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Principal Investigator, José Arturo Garrocho Rangel, Clinical Professor, Universidad Autonoma de San Luis Potosí
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U.A.S.L.P.; No funding (Other: No issuing organization)
Record Dates: First submitted 2025-11-27; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Local Anesthetic Infiltration; Topical Anesthesia; Pain Perception
Keywords: Topical dental anesthesia; Children; Anesthesia punction; Pain perception; Cryoanesthesia; Benzocaine
MeSH Terms: interventions — Anesthesia, Local; Lidocaine

STUDY DESIGN:
Intervention Model Description: A split-mouth randomized controlled clinical trial was conducted with 28 patients aged 6 to 12 years requiring bilateral inferior alveolar nerve blocks for bilateral lower arch dental treatment. Each participant received both anesthetic techniques in a randomized order on separate appointments, with treatment allocated to contralateral mandibular hemiarches. Primary and secondary outcome measures included pain intensity (Visual Analog Scale), heart rate, oxygen saturation, and behavioral response (FLACC scale).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryanesthesia. Topical anesthesia using application of ice cones, before anesthesic punction. (Experimental): Ice cones were prepared using sterile, individual-sized latex gloves filled with purified, sterile water. The open end of each glove was sealed and the glove was placed in a freezer (temperature: -18°C to -20°C) for minimum 24 hours prior to use. This produced a textured ice cone of approximately 5 cm × 3 cm suitable for direct application to the infiltration site.
  1. The application site (infiltration area on mucous membrane) was gently dried with sterile gauze.
  2. The ice cone was applied directly to the area using gentle circular rubbing motions.
  3. Duration of application: 60 seconds.
  4. Assessment: Observation for tissue blanching (white appearance) indicating adequate cooling.
  Interventions: Procedure: Local Anesthesia (lidocaine hydrochloride)
- Benzocaine group: Topical anesthesia using 20% benzocaine, before anesthetic punction. (Active Comparator): Benzocaine 20% Topical Anesthesia Technique:
  1. The application site was gently dried with sterile gauze
  2. Benzocaine 20% topical solution was applied using a sterile cotton applicator via gentle rubbing of the infiltration site
  3. Duration of application: 60 seconds
  4. No mechanical removal was performed; anesthetic was allowed to remain on tissue
  Interventions: Procedure: Local Anesthesia (lidocaine hydrochloride)

INTERVENTIONS:
Procedure: Local Anesthesia (lidocaine hydrochloride) — After topical anesthesia (either technique), the clinician proceeded with conventional inferior alveolar nerve block using standardized technique:
  1. Patient positioned recumbent in dental chair with mouth held open.
  2. Palpation of ipsilateral mandibular condyle by clinician's non-dominant hand.
  3. Cheek retracted with non-dominant hand to improve visualization.
  4. Long needle (27-gauge, 32 mm) inserted at horizontal level of contralateral mandibular canine, directed toward insertion of lateral pterygoid muscle below maxillary tuberosity.
  5. Needle advanced to contact medial mandibular wall (lingual surface).
  6. Aspiration performed to rule out intravascular needle placement.
  7. Injection of local anesthetic solution (1.8 mL of 2% lidocaine with 1:100,000 epinephrine).
  8. Needle carefully withdrawn following injection completion.
Procedure: Local Anesthesia (lidocaine hydrochloride) — After topical anesthesia (either technique), the clinician proceeded with conventional inferior alveolar nerve block using standardized technique:
  1. Patient positioned recumbent in dental chair with mouth held open
  2. Palpation of ipsilateral mandibular condyle by clinician's non-dominant hand
  3. Cheek retracted with non-dominant hand to improve visualization
  4. Long needle (27-gauge, 32 mm) inserted at horizontal level of contralateral mandibular canine, directed toward insertion of lateral pterygoid muscle below maxillary tuberosity
  5. Needle advanced to contact medial mandibular wall (lingual surface)
  6. Aspiration performed to rule out intravascular needle placement
  7. Injection of local anesthetic solution (1.8 mL of 2% lidocaine with 1:100,000 epinephrine)
  8. Needle carefully withdrawn following injection completion

SUMMARY:
This clinical study tested and compared two ways (cold-base technique or "cryoanesthesia" and conventional benzocaine gel) to reduce pain from dental injections in children.

Researchers worked with 28 children between 6 and 12 years old who needed injections on both sides of the lower jaw for dental treatment. Each child received cryoanesthesia on one side and 20% benzocaine gel on the other side, in different appointments, and the team measured pain, behavior, heart rate, and blood oxygen levels.

DETAILED DESCRIPTION:
Objective: To evaluate and compare pain perception during inferior alveolar nerve block puncture in pediatric patients using cryoanesthesia versus conventional topical benzocaine anesthesia.

Methods: A split-mouth randomized controlled clinical trial was conducted with 28 patients aged 6 to 12 years requiring bilateral inferior alveolar nerve blocks for bilateral lower arch dental treatment. Each participant received both anesthetic techniques in a randomized order on separate appointments, with treatment allocated to contralateral mandibular hemiarches. Primary and secondary outcome measures included pain intensity (Visual Analog Scale), heart rate, oxygen saturation, and behavioral response (FLACC scale).

ELIGIBILITY:
Inclusion Criteria:

* Systemic health: No significant medical history or uncontrolled systemic disease.
* Bilateral dental pathology requiring treatment: At least two teeth (one per mandibular hemiarch) requiring bilateral inferior alveolar nerve blocks for restorative or endodontic treatment.
* Cooperation level: Frankl behavioral rating scale classification III or IV (positive or very positive).
* Informed consent/Child assent: Signed informed consent from parent or legal guardian; signed assent from participant (age-appropriate).

Exclusion Criteria:

* Acute dental emergency requiring immediate treatment.
* Known hypersensitivity or allergy to benzocaine or other local anesthetics.
* Known hypersensitivity to cold (cryophobia or cold urticaria).
* Significant dental anxiety or phobia precluding study participation.
* Developmental delay or behavioral disorders limiting communication or cooperation.
* Current use of medications affecting pain perception or hemodynamic parameters.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Pain perception | Baseline: At the time of the anesthetic injection (or needle puncture) at the oral mucosa.
  Pain intensity was assessed using a validated instrument:
  Wong-Baker FACES® Pain Rating Scale (Visual Analog Scale): Immediately following completion of infiltration anesthesia injection, the participant was asked to indicate the level of pain experienced using the face scale (0 = no hurt to 10 = hurts worst).

SECONDARY OUTCOMES:
Heart Rate | Periprocedural: During the injection anesthetic procedure, from the anesthetic solution injection to the removal of the needle (approximately 45 seconds)
  Continuous pulse oximetry monitoring was conducted using a calibrated pulse oximeter (typical brands: Nellcor or equivalent) with appropriate pediatric finger probe or reusable sensor. Measurement unit: Pulses per minute (ppm) for heart rate (HR), which were recorded at two time points:
  1. Baseline measurement: Immediately before topical anesthetic application, with the participant in a calm resting state.
  2. During anesthetic infiltration: Recorded during active injection of local anesthetic solution into the infiltration site (oral mucosa).
Oxygen saturation | Periprocedural: During the injection anesthetic procedure, from the needle puncture to the removal of the needle (approximately 45 seconds).
  Percentage of blood's hemoglobin carrying oxygen (normally 95-100%). Continuous pulse oximetry monitoring was conducted using a calibrated pulse oximeter (typical brands: Nellcor or equivalent) with appropriate pediatric finger probe or reusable sensor. Measurement units: SpO2 percentage (%), which was recorded at two time points: 1. Baseline measurement: Immediately before topical anesthetic application, with the participant in a calm resting state. And 2. During infiltration measurement: During active injection of local anesthetic solution into the infiltration site.
Patient's behavioral response | Periprocedural: 45 seconds, from the anesthetic injection to the removal of the needle.
  Observable emotional and physiological reactions to the anesthetic injection through the FLACC (Facial expression, Legs, Activity, Cry, and Consolability) scale. Values: 0-10 (0 = relaxed, calm; 10 = severe distress).

CONTACTS AND LOCATIONS:
Overall Officials: Amaury Pozos Guillén, Ph.D., Study Director — Universidad Autónoma de San Luis Potosi
Locations (1):
- Pediatric Dentistry Postgraduate Program, Faculty of Denttistry, San Luis Potosí City, S.l.p., Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ninawe N, Anija CK. Comparative Evaluation of Effectiveness of Benzocaine Gel and Ice for Pain Management in Children during Local Anesthetic Administration by CCLAD: A Randomized Controlled Trial. Int J Clin Pediatr Dent. 2025 Jan;18(1):19-23. doi: 10.5005/jp-journals-10005-3045. Epub 2025 Feb 14. PMID 40110448
- [Background] Tirupathi SP, Rajasekhar S. Effect of precooling on pain during local anesthesia administration in children: a systematic review. J Dent Anesth Pain Med. 2020 Jun;20(3):119-127. doi: 10.17245/jdapm.2020.20.3.119. Epub 2020 Jun 24. PMID 32617406
- [Background] Lathwal G, Pandit IK, Gugnani N, Gupta M. Efficacy of Different Precooling Agents and Topical Anesthetics on the Pain Perception during Intraoral Injection: A Comparative Clinical Study. Int J Clin Pediatr Dent. 2015 May-Aug;8(2):119-22. doi: 10.5005/jp-journals-10005-1296. Epub 2015 Aug 11. PMID 26379379
- See also: Step-by-step instructions for performing oral cryotherapy — https://ostrowonline.usc.edu/oral-cryotherapy/